CLINICAL TRIAL: NCT00126165
Title: A Phase I/II Study of Escalated-dose Short-course Hypofractionated Radiotherapy (55 Gy/16 Fractions/4 Weeks) for Localized Prostate Cancer
Brief Title: Short-course Hypofractionated Radiotherapy for Localized Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alberta Health services (Other)
Collaborators: Calgary Health Region (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17885; 17885
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radiotherapy; hypofraction; radiosensitivity; image-guidance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: radiotherapy

SUMMARY:
This study is aimed at providing further clinical evidence to support or refute the current understanding of biological sensitivity of prostate cancer to fractionated radiotherapy. Determining the morbidity and cancer control provided by a 4-week course of treatment will greatly influence future radiotherapy services for patients with localized prostate cancer.

DETAILED DESCRIPTION:
This study is aimed at providing further clinical evidence to support or refute the current understanding of biological sensitivity of prostate cancer to fractionated radiotherapy. Determining the morbidity and cancer control provided by a 4-week course of treatment will greatly influence future radiotherapy services for patients with localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage T1 and T2 prostate cancer
* Prostate specific antigen (PSA)>=20 and Gleason score<=6
* PSA<=15 and Gleason score 7
* Signed informed consent

Exclusion Criteria:

* No hip prosthesis, pins or screws
* No previous pelvic radiotherapy
* No inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2004-09; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
rectal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Wu, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Wu JS, Brasher PM, El-Gayed A, Pervez N, Tai PT, Robinson J, Skarsgard D, Joseph K, Sia MA, Pearcey RG. Phase II study of hypofractionated image-guided radiotherapy for localized prostate cancer: outcomes of 55 Gy in 16 fractions at 3.4 Gy per fraction. Radiother Oncol. 2012 May;103(2):210-6. doi: 10.1016/j.radonc.2011.12.020. Epub 2012 Jan 24. PMID 22280805